CLINICAL TRIAL: NCT06384261
Title: Multicenter, Open-label, Randomized, Phase 2 Study of Venetoclax and Azacitidine Plus Cusatuzumab Versus Venetoclax and Azacitidine Alone in Newly Diagnosed AML Patients Who Are Not Candidates for Intensive Therapy
Brief Title: A Study Comparing Venetoclax and Azacitidine Plus Cusatuzumab to Venetoclax and Azacitidine in Newly Diagnosed AML Ineligible for Intensive Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OncoVerity, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OV-AML-1231
Record Dates: First submitted 2024-04-18; First posted 2024-04-25 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cusatuzumab in combination with venetoclax and azacitidine (Experimental): Cusatuzumab 20 mg/kg administered intravenously on days 3 and 17 in combination with venetoclax administered orally up to 400 mg once daily and azacitidine 75 mg/m^2 administered subcutaneously or intravenously once daily for 7 days of a 28 day cycle
  Interventions: Drug: Cusatuzumab; Drug: Venetoclax; Drug: Azacitidine
- Venetoclax in combination with azacitidine (Active Comparator): Venetoclax administered orally up to 400 mg once daily and azacitidine 75 mg/m^2 administered subcutaneously or intravenously once daily for 7 days of a 28 day cycle
  Interventions: Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Cusatuzumab — CD70 monoclonal antibody
  Other Names: OV-1001
  Arms: Cusatuzumab in combination with venetoclax and azacitidine
Drug: Venetoclax — BCL-2 inhibitor
Drug: Azacitidine — Hypomethylating agent

SUMMARY:
The goal of this clinical trial is to learn if participants treated with the experimental drug cusatuzumab added to venetoclax and azacitidine works to treat acute myeloid leukemia (AML) compared to venetoclax and azacitidine. Venetoclax and azacitidine are drugs commonly used to treat AML in patients that are unable to receive chemotherapy to treat AML. The main question the clinical trial aims to answer is does cusatuzumab added to venetoclax and azacitidine prolong the length of time participants live compared to venetoclax and azacitidine?

DETAILED DESCRIPTION:
This is a randomized, open-label, multicenter, Phase 2 trial to evaluate the efficacy, safety, and pharmacodynamics of cusatuzumab in combination with venetoclax and azacitidine compared to venetoclax and azacitidine in persons with newly diagnosed AML who are deemed ineligible for intensive chemotherapy.

Potential participants will be considered ineligible for intensive chemotherapy and, therefore, eligible for the study, if they meet the trial eligibility criteria and provide informed consent. Participants will undergo a diagnostic bone marrow biopsy and aspirate collected for pathology review, cytogenetics, fluorescence in situ hybridization (FISH), and polymerase chain reaction (PCR) analysis and other studies for confirmation of a diagnosis of AML and to define whether participants have adverse, intermediate, or favorable AML risk features. Participants will then be randomized 2:1 to either the experimental arm or the active comparator arm and stratified based on AML risk features (adverse, intermediate, and favorable risk).

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years old
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for the study and is willing to participate in the study
* Diagnosis of AML according to ICC 2022 (with the exclusion of MDS/AML with 10-19% blasts)
* Previously untreated AML except may have received emergency leukapheresis, hydroxyurea before study entry to control hyperleukocytosis
* Deemed unfit for intensive chemotherapy by meeting at least 1 of the following criteria:

  1. Participant is ≥75 years of age with Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 OR
  2. Participant is ≥18 to 74 years of age and has any of the following comorbidities:

     1. ECOG performance status of 2 or 3
     2. Cardiac status including any one of the following: congestive heart failure requiring treatment or ejection fraction ≤50% or chronic stable angina
     3. Known history of diffusion capacity of lung for carbon monoxide (DLCO) ≤65% of forced expiratory volume in the first second (FEV1) ≤65%
     4. Creatinine clearance (CrCl) ≥15 mL/min to <45 mL/min
     5. Hepatic disorder with total bilirubin >1.5 to 3x the upper limit of normal (ULN)
     6. Any other comorbidity that the investigators determine to be incompatible with conventional intensive chemotherapy
* Adequate liver and renal function defined as:

  1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <3xULN; for participants with leukemic infiltration of the liver (documented by biopsy or imaging), AST and ALT <5xULN is permitted
  2. Total bilirubin ≤1.5xULN, unless bilirubin rise is due to Gilbert's syndrome or of nonhepatic origin. Participants who are <75 years of age may have a bilirubin up to 3xULN.
  3. Estimated glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2 (by the Modification of Diet in Renal Disease [MDRD] formula). Participants who are <75 years of age may have an eGFR ≥15 mL/min/1.73 m2.
* Women of childbearing potential (WOCBP), defined as fertile women between menarche and post menopause unless permanently sterile, must have a negative highly sensitive serum β-human chorionic gonadotropin (β-hCG) or urine pregnancy test at screening
* Must be willing to use contraception as consistent with institutional guidelines regarding the use of contraceptive methods for participants participating in clinical studies

  1. WOCBP must agree to adhere to the following birth control measures while receiving study treatment continuing to 3 months after the last dose of study drug:

     1. Must be practicing a highly effective method of birth control (failure rate of <1% per year when used consistently and correctly) as determined by institutional standards
     2. Must agree to not donate eggs (ova, oocytes) for the purposes of assisted reproduction
     3. Must not be breastfeeding and not planning to become pregnant
  2. Male participants who are sexually active with WOCBP, and male partners of study participants who are WOCBP, and who are not surgically or otherwise sterile must agree to adhere to the following birth control measures while receiving study treatment and for 3 months after the last dose of study drug:

     1. Must agree to use a barrier method of birth control (e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap [diaphragm or cervical/vault caps] with spermicidal foam, gel, film, cream, or suppository)
     2. Must not donate sperm
     3. Must no plan to father a child
* Participants with HIV infection are eligible for the trial if the following criteria are met:

  1. CD4+ T-cell count ≥200 cells/μL
  2. No prior history of AIDS-defining opportunistic infection within the past 12 months
  3. Receiving treatment with antiretroviral therapy
  4. Undetectable viral load within 6 months of screening

Exclusion Criteria:

* Any prior treatment for AML (except those outlined in inclusion criterion #4)
* Participant has received a hypomethylating agent (HMA) or venetoclax for MDS or myeloproliferative neoplasm
* Leukemic involvement in the central nervous system
* Participants with acute promyelocytic leukemia (APL)
* ECOG performance status of 4 for participants 18 to 74 years of age and ECOG performance status of 3 or 4 for participants ≥75 years of age
* Use of immune suppressive agents ≤4 weeks before the first administration of cusatuzumab. Participants may be included if free of systemic corticosteroids >5 days before the first administration of cusatuzumab with the exception of corticosteroids at physiologic replacement doses.
* Received a live, attenuated vaccine within 4 weeks prior to initiation of study drug
* Active malignancies (i.e., progressing or requiring treatment change in the last 24 months) other than the disease being treated under study. Exceptions to this exclusion criterion include the following:

  1. Nonmelanoma skin cancer treated within the last 24 months that is considered completely cured
  2. Adequately treated breast lobular carcinoma in situ and breast ductal carcinoma in situ
  3. Adequately treated cervical carcinoma in situ and breast ductal carcinoma in situ
  4. History of localized breast cancer and receiving anti-hormonal agents, or history of localized prostate cancer (N0M0) and receiving androgen depravation therapy
  5. A malignancy that is considered cured with minimal risk of recurrence
* Any active systemic infection
* History of prior HSCT (allogeneic or autologous transplants)
* Active hepatitis B or C infection or other clinically active liver diseases ad defined below:

  1. Seropositivity for hepatitis B is defined by a positive test for hepatitis B surface antigen (HBsAg)
  2. Participants with resolved infection (i.e., participants who are HBsAg negative with antibodies to total hepatitis B core antigen [anti-HBc] with or without the presence of hepatitis B surface antibody [anti-HBs]) must be screened using PCR measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded.

     * Participants with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR
  3. Active hepatitis C infection as defined by being positive for a nucleic acid test for hepatitis C virus (HCV) RNA
* Congestive hear failure severity that is New York Heart Association Class III or IV
* Unstable angina
* Known allergies, hypersensitivity, or intolerance to cusatuzumab, venetoclax, or azacitidine or their excipients (e.g., mannitol, an excipient of azacitidine)
* Inability or difficulty swallowing capsules/tablets, malabsorption syndrome, or any disease or medical condition significantly affecting gastrointestinal function
* Any condition for which, in the investigator's opinion, participation would not be in the best interest of the participant (e.g., compromise the well-being) or physical limitations that could prevent, limit, or confound the protocol-specified assessments
* Major surgery (e.g., requiring general anesthesia) ≤4 weeks prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause, assessed up to 5 years
  In all randomized participants

SECONDARY OUTCOMES:
Complete Remission rate (CR) | From date of randomization to relapse or criteria for refractory disease are met, assessed up to 3 years
  Proportion of participants achieving CR per the European LeukemiaNet (ELN) 2022 criteria
Event-free survival (EFS) | From date of randomization to date of treatment failure, hematologic relapse from CR/CRh/CRi or death from any cause, assessed up to 5 years
  Defined per ELN 2022 criteria
Composite CR rate (CRc) | From date of randomization to relapse or criteria for refractory disease are met, assessed up to 3 years
  Sum of CR+CRh+CRi rate. CRh is defined as CR with partial hematologic recovery. CRi is defined as CR with incomplete hematologic recovery. Defined per ELN 2022 criteria.
Rate of CRh and CRi | From date of randomization to relapse or criteria for refractory disease are met, assessed up to 3 years
  Defined per ELN 2022 criteria
Duration of CR | From date of first CR to hematological relapse or death from any cause, assessed up to 5 years
  Defined per ELN 2022 criteria
Time to first CR | From date of randomization to first occurrence of CR, assessed up to 3 years
  Defined per ELN 2022 criteria
Rate of minimal residual disease (MRD) negativity in patients achieving CR, CRh, or CRi | From date of randomization to relapse or criteria for refractory disease are met, assessed up to 5 years
  Defined per ELN 2022 criteria and guidelines for testing
Proportion of participants proceeding to hematopoietic stem cell transplantation (HSCT) | From date of randomization to date of HSCT, assessed up to 5 years
OS in participants undergoing HSCT | From date of randomization to death from any cause, assessed up to 5 years
Incidence of adverse events (AEs), serious adverse events (SAEs), and AEs leading to study drug discontinuation | Signing of informed consent to 30 days after the last dose of study treatment or until start of subsequent anti-AML therapy
  Per CTCAE criteria
Incidence of dose modifications due to AEs | Randomization to 30 days after the last dose of study treatment or until start of subsequent anti-AML therapy
  Includes interruptions and/or delays
Number of participants with abnormal laboratory test results | Signing of informed consent to 30 days after the last dose of study treatment or until start of subsequent anti-AML therapy
  Findings will be summarized
Incidence of anti-drug antibodies (ADA) and neutralizing antibodies (NAb) | From date of randomization to end of treatment, assessed up to 5 years
Overall survival in subgroups of participants according to specified AML risk stratification models | From date of randomization to death from any cause, assessed up to 5 years
Complete Remission rate | From date of randomization to relapse or criteria for refractory disease are met, assessed up to 3 years
  In subgroups of participants according to specified AML risk stratification models. CR defined per ELN 2022 criteria.

CONTACTS AND LOCATIONS:
Locations (31):
- United States (17):
  - Banner MD Anderson, Gilbert, Arizona
  - City of Hope, Duarte, California
  - University of California Los Angeles, Los Angeles, California
  - University of Colorado Health - Anschutz Cancer Pavilion - Anschutz Medical Campus, Aurora, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - AdventHealth Medical Group Blood & Marrow Transplant at Orlando, Orlando, Florida
  - The University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Norton Healthcare, Inc., Louisville, Kentucky
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Hofstra/Northwell Health, Lake Success, New York
  - Cornell University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Wake Forest North Carolina, Winston-Salem, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Fred Hutch Seattle Cancer Care Alliance, Seattle, Washington
  - Medical College of Wisonsin, Milwaukee, Wisconsin
- Canada (7):
  - Tom Baker Cancer Center-Alberta Health Services - University of Calgary, Calgary, Alberta
  - Stollery Children's Hospital-Walter C Mackenzie Health Sciences Centre - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - University of Western Ontario, London, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Saskatchewan Cancer Agency - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Germany (4):
  - Marien Hospital Duesseldorf, Düsseldorf
  - Universitaetsklinik Frankfurt, Frankfurt
  - Medizinische Hochschule Hanover, Hannover Medical School, Hanover
  - Universitaetsklinik um Schleswig-Holstein, UKSH-Campus Kiel, Kiel
- Switzerland (3):
  - Inselspital Bern, Bern
  - HFR Fribourg - Hopital Cantonal, Fribourg
  - Kantonsspital St. Gallen, Sankt Gallen